CLINICAL TRIAL: NCT04450641
Title: A Gamified Mobile Platform for Improving Social Communication in Children With Autism
Brief Title: Piloting a Mobile Game for Behavioral Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Dennis Paul Wall, Associate Professor, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 39562
Record Dates: First submitted 2020-06-24; First posted 2020-06-29 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: digital; mobile health; game; autism; technology; therapy
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: All participants who complete baseline measures will be directed to download the GuessWhat app. Participants who do not download the GuessWhat app and elect not to play, will be assigned to the Inactive Users group during analysis.
Masking Description: No masking. All participants received the same condition and asked to play a mobile app. Participants who did not play the app during piloting were asked to complete study measures pre and post. These measures were compared against participants who did play the app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Treatment group used GuessWhat during the 4 week intervention period.
  Interventions: Other: GuessWhat Mobile Application
- Control (Other): Participants in control group received standard treatment as usual.
  Interventions: Other: GuessWhat Mobile Application

INTERVENTIONS:
Other: GuessWhat Mobile Application — The GuessWhat app is a charades style game and app that engages parent and child in fluid social interaction where the parent must guess what the child is acting out based on the prompt shown on the phone screen. Participants will use their own personal phone to download the study app. Parent and child will be encouraged to play using the emojis and emotion game mode at least 3 individual game sessions per week. Parents are asked to play GuessWhat with their child 3-4 times per week for 4 weeks.

SUMMARY:
The following study aims to understand the feasibility of the mobile app and game, GuessWhat, to deliver behavioral therapy to children with autism. The GuessWhat app is a charades style game that engages parent and child in fluid social interaction where the parent must guess what the child is acting out based on the prompt shown on the phone screen. Participants will use their own personal phone to download the study app. The app will walk participants through a variety of charades style games. The interactive games will be video recorded and all data are transferred securely to the Wall Lab for analysis. This study is enrolling parents of children with ASD who are at least 18 years of age and have a child between 3-12 years old. Parents are asked to complete questionnaires before and after playing the GuessWhat game with their child 3-4 times per week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Parent who is at least 18 years old of child with autism.
* Child with autism is between 3 and 12 years old at time of baseline data collection.

Exclusion Criteria:

* Parent is not able to read or speak English
* Parent does not have an Android or iOs smartphone compatible with GuessWhat App

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in parent reported social responsiveness from week 0 to week 4 | Baseline (Week 0), Week 4
  The Social Responsiveness Scale-2 is a 65-item measure where parents rate their child selecting responses on a Likert Scale. This measure will be used to measure and identify social impairment associated with Autism Spectrum Disorder (ASD) and to quantify its severitySocial Responsiveness Scale (SRS) raw scores measure social abilities with lower scores indicating better social skills. (Raw Score Range: 0 - 195 and T-Score Range: 37- above 90).
Change in parent reported socialization subscale scores of the Vineland Adaptive Behavior Scales,2nd Edition (VABS-II) from baseline to week 4 | Baseline (Week 0), Week 4
  Vineland Adaptive Behavior Scales, 2nd edition (VABS-II) Socialization subscale of the Parent/Caregiver Comprehensive form will be administered online to the parents. Scores from the socialization domain of the VABS-III reflects one's functioning in social situations. The socialization subscale is 32 items, where raw scores are converted to IQ-type standard scores--v-scale scores (M=15, SD=3) where scores range from 1 to 24, and factor in age equivalents, growth scale values, and higher scores indicate better adaptive functioning.

SECONDARY OUTCOMES:
GuessWhat App Usage Data | 4 weeks
  App usage data comprised of game decks selected, number of game sessions started, ended, and shared.
Parent reported feedback | Week 4
  Qualitative survey delivered to parent participants at Week 4 to understand preferred games, overall feedback including likes and dislikes, any technical issues they experienced or challenges in using the app.
Change in parent reported communication subscale scores of the Vineland Adaptive Behavior Scales,2nd Edition (VABS-II) from baseline to week 4 | Baseline (Week 0), Week 4
  Vineland Adaptive Behavior Scales, 2nd edition (VABS-II) Communication subscale of the Parent/Caregiver Comprehensive form will be administered online to the parents. Scores from the communication domain of the VABS-III reflects The communication subscale is 32 items, where raw scores are converted to IQ-type standard scores--v-scale scores (M=15, SD=3) where scores range from 1 to 24, and factor in age equivalents, growth scale values, and higher scores indicate better adaptive functioning.

OTHER OUTCOMES:
Baseline Parent Reported Social Communication | Baseline (Week 0)
  The Social Communication Questionnaire (SCQ) screens for autism in children over 4:0 years in age. Parents are asked 40 Yes/No questions and the resulting score is out of 39 (the first question is not associated with a numerical value). The SCQ assesses a child's communication skills and social functioning. It takes less than 10 minutes to complete and is administered by clinical research coordinators to parents of children during the phone screen to participants who have already completed the online screening questionnaire. A score of 15 or above is indicative of autism and is required to be eligible in the research study.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Wall, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Website — http://guesswhat.stanford.edu